CLINICAL TRIAL: NCT05572671
Title: Linking Brain Network Dynamics to Imminent Smoking Lapse Risk and Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Stephen Wilson, Associate Professor of Psychology, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00020857
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use

STUDY DESIGN:
Intervention Model Description: Participants will complete a task (the behavioral intervention) designed to model smoking lapse behavior in the laboratory; during the task, they will be given the option of delaying smoking in exchange for monetary reinforcement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fMRI smoking lapse task (Experimental)
  Interventions: Behavioral: Laboratory task modeling smoking lapse behavior

INTERVENTIONS:
Behavioral: Laboratory task modeling smoking lapse behavior — Participants will complete a task (the behavioral intervention) designed to model smoking lapse behavior in the laboratory; during the task, they will be given the option of delaying smoking in exchange for monetary reinforcement.

SUMMARY:
Most attempts to quit smoking end in relapse, or a return to regular smoking. One of the biggest threats to cessation is a lapse (i.e., any cigarette use during a quit attempt). Thus, characterizing why lapses occur is essential to understanding and preventing smoking relapse. Functional magnetic resonance imaging (fMRI) is a promising method for characterizing the psychological processes that lead to smoking lapses because it provides a way to measures patterns of brain activity thought to reflect relevant mental processes as they change over time. However, methodological issues have hindered the ability to capitalize on this potential and prevented an understanding of how brain activity and corresponding psychological processes unfold in the critical moments that immediately precede a smoking lapse. The proposed project will address this knowledge gap using a novel fMRI paradigm adapted from a well-validated behavioral lapse task. The goals of the project are to characterize changes in brain activity that lead up to a lapse and to investigate how these changes are related to concurrent affect and subsequent cigarette use.

DETAILED DESCRIPTION:
Most attempts to quit smoking end in relapse, or a return to regular smoking. One of the biggest threats to cessation is a lapse (i.e., any cigarette use during a quit attempt). Thus, characterizing why lapses occur is essential to understanding and preventing smoking relapse. Functional magnetic resonance imaging (fMRI) is a promising method for characterizing the psychological processes that lead to smoking lapses because it provides a way to measures patterns of brain activity thought to reflect relevant mental processes as they change over time. However, methodological issues have hindered the ability to capitalize on this potential and prevented an understanding of how brain activity and corresponding psychological processes unfold in the critical moments that immediately precede a smoking lapse. The proposed project will address this knowledge gap using a novel fMRI paradigm adapted from a well-validated behavioral lapse task. This novel fMRI paradigm includes an in-scanner delay period that models the ability to resist smoking during acute nicotine abstinence and a post-scan ad-lib period that captures key aspects of the smoking behavior that follows. Adults who smoke will abstain from cigarettes for 12 hours before completing the fMRI lapse paradigm. The goals of the project are to characterize changes in brain activity that lead up to a lapse and to investigate how these changes are related to concurrent affect and subsequent cigarette use. The study will focus specifically on linking lapse-related outcomes to time-dependent interactions between two large-scale brain networks: the executive control network, which includes parts of the lateral prefrontal and parietal cortices, and the default mode network, which includes parts of the medial prefrontal and posterior cingulate cortices. The central hypothesis guiding the proposed research is that lapse-related behavior and affect will be predicted by the extent to which the default mode network and the executive control network are functionally segregated (i.e., the strength of the connectivity within the default mode and executive control networks, relative to connectivity between the networks). The aims of the project are: 1) To examine the association between time-dependent changes in brain network dynamics and subsequent risk of smoking lapse; 2) To examine the association between time-dependent changes in brain network dynamics and self-reported affect leading up to a smoking lapse; and 3) To examine the association between brain network dynamics directly before a lapse and reinforcement from the smoking that follows. An additional exploratory aim of the study is to evaluate potential moderators of the association between brain network dynamics and lapse-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 21 and 65.
* Participants must be fluent English speakers.
* Participants must pass an MRI safety screening.
* Participants must report smoking at least six cigarettes per day continuously for at least the 12 preceding months.
* Participants must have a baseline expired-air carbon monoxide exceeding 10 parts per million in order to verify smoking status.

Exclusion Criteria:

* Individuals will be excluded if they report that they are not willing to refrain from using nicotine for 12 hours before the experimental lab visit.
* Individuals will be excluded if they have any known risk from exposure to high-field strength magnetic fields (e.g., pacemakers), any irremovable metallic foreign objects in their body (e.g., braces), or a questionable history of metallic fragments that are likely to create artifact on the MRI scans.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Blood-oxygen-level dependent (BOLD) signal | Day 2 (Visit 2)
  Blood-oxygen-level dependent (BOLD) signal measured using functional magnetic resonance imaging
Self-reported affect | Day 2 (Visit 2)
  Self-report ratings of affective valence and arousal

SECONDARY OUTCOMES:
Self-reported craving and nicotine withdrawal symptoms | Day 2 (Visit 2)
  Self-report ratings of level of craving and other common nicotine withdrawal symptoms (e.g., irritability)

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided